CLINICAL TRIAL: NCT00541515
Title: Closing the Loop Between Glucose Sensor and Insulin Pump-developing an Algorithm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: rmc004706ctil
Record Dates: First submitted 2007-10-08; First posted 2007-10-10 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-04

CONDITIONS: Diabetes, Type I
Keywords: Type 1 diabetes; Artificial pancreas; Insulin Pump
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- closed loop system (Experimental): Device: continuous glucose sensors and insulin pump
  Interventions: Device: continuous glucose sensors and insulin pump

INTERVENTIONS:
Device: continuous glucose sensors and insulin pump — continuous glucose sensors and insulin pump

SUMMARY:
An open interventional data collection study in order to build a database to close the loop between glucose sensor and insulin pump.

background: The ultimate goal in diabetes treatment is to develop an autonomous insulin delivery system (artificial pancreas) capable of continuous glucose sensing, thereby mimicking the physiologic function of the islet beta cells and freeing the patient from the need for constant calculations of daily insulin and carbohydrates. Several prototypes of closed-loop system have been developed in recent years, based on different types of control algorithms, to establish the connection between the sensor and the insulin pump. Current research in the formulation of this type of subcutaneous closed-loop system still faces major challenges, therefore, there is a need for further study and evaluation.

Objectives:

1. To evaluate the lag time of the effect of subcutaneous insulin infusion on blood glucose levels by using continuous glucose sensor
2. To measure the insulin sensitivity as expressed by changes in blood glucose levels after s.c insulin infusion .
3. To evaluate real time sensor calibration algorithms based on the measured lag times
4. Collecting clinical data in order to develop and evaluate mathematical models which will serve a base to simulators.
5. Developing and accessing advanced learning and control algorithms as a step towards developing an artificial pancreas

ELIGIBILITY:
Inclusion Criteria:

1. Diabetes type 1 for at least one year.
2. ages >10 years.
3. signed informed consent form.
4. willing to cooperate with all study requirements.

Exclusion Criteria:

1. Sensor allergy.
2. Psychiatrist diseases.
3. other chronic diseases.
4. Participation in another study that involves a medicine or a medical device.Subjects have to finish participating in other studies at least 30 days before joining this study. Each subject can participate in this study only once.

Ages: 10 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2007-10; Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Blood glucose levels | countinuasly

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Phillip, Professor, Principal Investigator — Schneider Children Medical Center
Locations (1):
- schneider children medical center of Israel, Petah Tikva, Israel

REFERENCES:
- [Derived] Nimri R, Atlas E, Ajzensztejn M, Miller S, Oron T, Phillip M. Feasibility study of automated overnight closed-loop glucose control under MD-logic artificial pancreas in patients with type 1 diabetes: the DREAM Project. Diabetes Technol Ther. 2012 Aug;14(8):728-35. doi: 10.1089/dia.2012.0004. PMID 22853723
- [Derived] Atlas E, Nimri R, Miller S, Grunberg EA, Phillip M. MD-logic artificial pancreas system: a pilot study in adults with type 1 diabetes. Diabetes Care. 2010 May;33(5):1072-6. doi: 10.2337/dc09-1830. Epub 2010 Feb 11. PMID 20150292